CLINICAL TRIAL: NCT02184468
Title: Dual Dispatch of EMS, Fire Fighters and/or Police in Out-of-hospital Cardiac Arrest Implemented in Nine Counties in Sweden - Can More Lives be Saved by Using This Method?
Brief Title: Survival Study After Out-of-hospital Cardiac Arrest
Acronym: SAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Laerdal Foundation (Other); Swedish Heart Lung Foundation (Other); Ministry of Health and Social Affairs, Sweden (Other Government); Swedish Association of Local Authorities and Regions (Other)
Responsible Party: Principal Investigator, Leif Svensson, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SAMS 242-11
Record Dates: First submitted 2014-06-27; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Cardiac Arrest; Out-of-Hospital Cardiac Arrest; Firefighters; Police; Defibrillators; Survival
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dual dispatch (Other): Simultaneously dispatching of EMS, firefighters and/or police in OHCA
  Interventions: Other: Simultaneously dispatch of firefighters and/or police in case of OHCA

INTERVENTIONS:
Other: Simultaneously dispatch of firefighters and/or police in case of OHCA — In case of OHCA, firefighters and/or police trained in CPR and equipped with AEDs will be dispatched in parallel with EMS in nine counties in Sweden.

SUMMARY:
The purpose of this study is to determine if dual dispatch of ambulance, fire fighters and/or police in out-of-hospital cardiac arrest (OHCA), can reduce the time to cardiopulmonary resuscitation (CPR) and defibrillation, thus increasing survival.

DETAILED DESCRIPTION:
Hypothesis If simultaneous dispatch of ambulance (EMS), firefighters and/or police is being initiated when an OHCA occurs, then the two latter units will be first at scene, before the ambulance crew, in ≥30% of the cases. We anticipate therefore that overall 30-days survival will increase on a national level from 9% to 12%.

Method During the period 110901 to 141231 all OHCA cases will be analyzed were the emergency medical communication centre (EMCC) has dispatched ambulance, firefighters and/or the police. Participating in the Saving More Lives in Sweden (SAMS) project are the following counties: Stockholm, Sodermanland, Jonkoping, Vastra Gotaland (VG Region), Halland, Dalarna, Jamtland, Kalmar and Uppsala. Data is collected by the units being dispatched and thereafter sent on line to a database managed by Registercentrum in Gothenburg (http://www.registercentrum.se/), administrators of the Swedish Cardiac Arrest Register.

Parameters obtained are:

* Time for dispatch of fire fighters and/or police (recorded digitally).
* Time for arrival to the patient.
* Verification if cardiac arrest or not.
* CPR performed by fire fighters or police before arrival of EMS.
* Automated External Defibrillator (AED) connected to the patient.
* If yes, was the first recorded rhythm shockable, i.e. ventricular fibrillation (VF) or pulseless ventricular tachycardia (VT).
* Time to defibrillation.

Survival data during from the Swedish Cardiac Arrest Register (SCAR) will be obtained during the same time period from nine comparable Swedish regions not participating in the SAMS study.

ELIGIBILITY:
Inclusion Criteria:

* All cases where the dispatcher suspects cardiac arrest, i.e. unconscious person with abnormal or no breathing

Exclusion Criteria:

* Children < 8 y
* Obviously deceased persons according to regulations in EMS protocols

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 30-days after out-of-hospital cardiac arrest (OHCA)

SECONDARY OUTCOMES:
Time for dispatching of fire fighters and/or police | Up to 1 y after ending recruitement
  Data are obtained digitally from the dispatch center.
Time for arrival to the patient | Up to 1 y after ending recruitement
  Data are collected both digitally from the dispatch center and from protocols sent in on line by first responders.
Time for attaching the defibrillator to the patient | Up to 1 y after ending recruitement
  Data are collected from protocols sent in on line by first responders.
Time to first defibrillation | Up to 1 y after ending recruitement
  Data collected from the protocol sent in on line by first responders.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Svensson, MD, PhD, Principal Investigator — Center for Resuscitation Science, Karolinska Institutet, Stockholm, Sweden
Locations (1):
- Center for Resuscitation Science, Sodersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Hasselqvist-Ax I, Nordberg P, Herlitz J, Svensson L, Jonsson M, Lindqvist J, Ringh M, Claesson A, Bjorklund J, Andersson JO, Ericson C, Lindblad P, Engerstrom L, Rosenqvist M, Hollenberg J. Dispatch of Firefighters and Police Officers in Out-of-Hospital Cardiac Arrest: A Nationwide Prospective Cohort Trial Using Propensity Score Analysis. J Am Heart Assoc. 2017 Oct 4;6(10):e005873. doi: 10.1161/JAHA.117.005873. PMID 28978527